CLINICAL TRIAL: NCT00801762
Title: Fiber-Optic Confocal Microscopy of the Urinary Tract Histopathology
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: Mauna Kea Technologies (Industry)
Other Study IDs: SU-10142008-1319
Record Dates: First submitted 2008-12-02; First posted 2008-12-03 (Estimated); Last update posted 2019-04-22 (Actual); Status verified 2019-04

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Device: Fibered confocal microscope

SUMMARY:
The goal of the study is to develop a novel approach to obtain real time optical biopsy of urinary tract pathology (e.g., bladder tumors) during urinary tract endoscopy using a novel fibered confocal microscope.

ELIGIBILITY:
Inclusion Criteria:Research subjects with suspected urinary tract pathology (e.g., bladder tumors) who are scheduled to undergo cystoscopy with possible excisional biopsy (e.g. transurethral resection of bladder tumor) in the operating room.
 Exclusion Criteria:History of hypersensitivity to fluorescein; active urinary tract infection; pregnant; currently breast feeding;

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2008-09 (Actual); Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph C. Liao, Principal Investigator — Stanford University
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, California, United States

REFERENCES:
- [Derived] Sonn GA, Jones SN, Tarin TV, Du CB, Mach KE, Jensen KC, Liao JC. Optical biopsy of human bladder neoplasia with in vivo confocal laser endomicroscopy. J Urol. 2009 Oct;182(4):1299-305. doi: 10.1016/j.juro.2009.06.039. Epub 2009 Aug 14. PMID 19683270